CLINICAL TRIAL: NCT06760624
Title: Effectiveness of Ofatumumab in Real-world Practice
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157AUS21
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Ofatumumab MS Cohort: Adult patients diagnosed with MS who were treated with ofatumumab.
- Anti-CD20-naïve Sub-cohort: Adult patients diagnosed with MS who were treated with ofatumumab and had not received anti-CD20 treatment.
- Anti-CD20-experienced Sub-cohort: Adult patients diagnosed with MS who were treated with ofatumumab and had previously received anti-CD20 treatment.

SUMMARY:
This study used a retrospective single cohort pre-post design on Optum® Clinformatics® Data Mart (CDM) data from 20 August 2019 to 31 December 2023 (study period). Patients with a diagnosis of multiple sclerosis (MS) treated with ofatumumab (OMB) between 20 August 2020 (U.S. Food and Drug Administration [FDA] approval date) and 01 July 2023 (patient identification window) were included in the study population. The date of the first OMB claim within the patient identification window was defined as the index date. Outcomes, including annualized relapse rate (ARR) and MS-related healthcare resource utilization (HCRU), were measured across two distinct periods. The pre-index period was defined as the fixed 12-month period prior to the index date, during which demographic and clinical characteristics were also assessed. The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another disease modifying therapy [DMT]), discontinuation of enrollment, or end of study period on 31 December 2023.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 years or older as of the index date corresponding to the initial claim for OMB therapy.
2. One claim or more for OMB therapy recorded during the patient identification period (index date = date of the first claim for OMB).
3. One claim or more with a diagnosis of MS (International Classification of Diseases, Tenth Revision [ICD-10] code G35.xx) any time before the index date and up to 6 months after the index date.
4. Continuous healthcare plan enrollment from ≥12 months prior to the index date (pre-index period) to ≥12 months following the index date (post-index period).
5. Persistent use of OMB therapy throughout the post-index period, defined as the absence of a discontinuation of OMB or switch to another MS treatment.

Exclusion criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 779 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) in the Pre-Index Period | 12 months
  The pre-index period was defined as the fixed 12-month period prior to the index date. The index date was the date of the first OMB claim. The ARR was defined as the number of relapse events per person-year.
ARR in the Post-index Period | An average of approximately 16 months
  The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another disease modifying therapy [DMT]), discontinuation of enrollment, or end of study period. The index date was the date of the first OMB claim. The ARR was defined as the number of relapse events per person-year.
Incidence Rate Ratio | An average of approximately 16 months
  Incidence rate ratio was measured to evaluate the change in MS-related ARR in the pre- versus the post-index period.
  The index date was the date of the first OMB claim. The pre-index period was defined as the fixed 12-month period prior to the index date. The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period.

SECONDARY OUTCOMES:
Age | Baseline
Number of Patients per Demographic Category | Baseline
  Demographic categories included:
  * Age Group (18-34, 35-44, 45-54, 55-64, and 65+ years)
  * Gender
  * Race
  * Region
  * Insurance Payer type
  * Year of Index date (2020, 2021, 2022)
Mean Deyo-Charlson Comorbidity Index | Baseline
  Deyo-Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions. Comorbidity was assessed using the Charlson Comorbidity Index (CCI), categorized as low (0-1) and high (≥2).
Mean Number of Psychiatric Diagnostic Group (PDG) Mental Health Disorders | Baseline
  PDG captures a list of mental health disorders a patient may have at study baseline. The following are the list of PDGs:
  * Adult personality disorders
  * Anxiety disorders
  * Behavioral syndromes
  * Childhood and adolescent psychiatric syndromes
  * Intellectual disabilities
  * Psychiatric disorders with known physiological causes
  * Mood disorders
  * Pervasive disorders
  * Schizophrenia
  * Substance use
Number of Patients Categorized by Top Five Selected Comorbidities | Baseline
  Top five selected comorbidities included osteoarthritis, dyslipidemia, depression, hypertension, and sleep disorders.
Number of Patients Categorized by Top Five MS-related Symptoms and Secondary Conditions | Baseline
  Top five MS-related symptoms and secondary conditions included anxiety, fatigue or malaise, sensory problems, eye symptoms, and urinary tract infection.
Number of Patients Categorized by MS Disability Level | Baseline
  MS disability level was based on observance of Expanded Disability Status Scale (EDSS)-related symptoms and durable medical equipment (DME) use observed in claims data weighted by severity score. Disability levels and definitions were as follows: Severe = Defined as having ≥1 EDSS-related symptom with severity score = 3 in any functional system; Moderate: Defined as having ≥1 EDSS-related symptom with severity score = 2 in any functional system, or having ≥2 functional systems with severity score = 1; Mild: Defined as having only one EDSS-related symptom with severity score = 1 or having no EDSS-related symptoms observed during the measurement period.
Number of Patients Categorized by DMT Used in the Pre-index Period | Baseline
  DMT categories included:
  * Any DMT
  * Low/moderate efficacy therapy
  * High efficacy therapy
  * No DMT
Pre-index Healthcare Resource Utilization (HCRU): Number of MS-related Hospitalizations per Person-year (PPY) | 12 months
  The pre-index period was defined as the fixed 12-month period prior to the index date. The index date was the date of the first OMB claim.
Pre-index HCRU: Number of Days of MS-related Hospitalization PPY | 12 months
  The pre-index period was defined as the fixed 12-month period prior to the index date. The index date was the date of the first OMB claim.
Pre-index HCRU: Number of MS-related Healthcare Visits PPY | 12 months
  The pre-index period was defined as the fixed 12-month period prior to the index date. The index date was the date of the first OMB claim. MS-related healthcare visits included emergency department visits and outpatient visits.
Post-index HCRU: Number of MS-related Hospitalizations PPY | An average of approximately 16 months
  The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period. The index date was the date of the first OMB claim.
Post-index HCRU: Number of Days of MS-related Hospitalization PPY | An average of approximately 16 months
  The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period. The index date was the date of the first OMB claim.
Post-index HCRU: Number of MS-related Healthcare Visits PPY | An average of approximately 16 months
  The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period. The index date was the date of the first OMB claim. MS-related healthcare visits included emergency department visits and outpatient visits.
Incidence Rate Ratio of MS-related Hospitalizations | An average of approximately 16 months
  Incidence rate ratio was measured to evaluate the change in MS-related hospitalizations in the pre- versus the post-index period.
  The index date was the date of the first OMB claim. The pre-index period was defined as the fixed 12-month period prior to the index date. The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period.
Incidence Rate Ratio of Days of MS-related Hospitalizations | An average of approximately 16 months
  Incidence rate ratio was measured to evaluate the change in days of MS-related hospitalizations in the pre- versus the post-index period.
  The index date was the date of the first OMB claim. The pre-index period was defined as the fixed 12-month period prior to the index date. The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period.
Incidence Rate Ratio of MS-related Emergency Department Visits | An average of approximately 16 months
  Incidence rate ratio was measured to evaluate the change in MS-related emergency department visits in the pre- versus the post-index period.
  The index date was the date of the first OMB claim. The pre-index period was defined as the fixed 12-month period prior to the index date. The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period.
Incidence Rate Ratio of MS-related Outpatient Visits | An average of approximately 16 months
  Incidence rate ratio was measured to evaluate the change in MS-related outpatient visits in the pre- versus the post-index period.
  The index date was the date of the first OMB claim. The pre-index period was defined as the fixed 12-month period prior to the index date. The post-index period was defined as the variable period of ≥6 months after the index date, extending until the earliest between the end of persistent OMB use (defined as last day of OMB supply before a gap of ≥60 days or switch to another DMT), discontinuation of enrollment, or end of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for COMB157AUS21 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18261